CLINICAL TRIAL: NCT06167655
Title: A PIVOTAL STUDY EVALUATING SAFETY AND EFFICACY OF THE SHIRATRONICS MIGRAINE THERAPY SYSTEM IN RELIEVING, INTERRUPTING, AND PREVENTING CHRONIC MIGRAINE (RELIEV-CM2)
Brief Title: A PIVOTAL STUDY EVALUATING SAFETY AND EFFICACY OF THE SHIRATRONICS MIGRAINE THERAPY SYSTEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ShiraTronics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STCM02
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Headache Migraine Chronic
MeSH Terms: interventions — Implantable Neurostimulators

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- High Dose (Active Comparator)
  Interventions: Device: Neurostimulator
- Low Dose (Sham Comparator)
  Interventions: Device: Neurostimulator

INTERVENTIONS:
Device: Neurostimulator — Neurostimulation system that applies stimulation to nerve pathways in the head associated with migraine symptoms.

SUMMARY:
Prospective, multi-center, double blind, randomized, sham-controlled study to evaluate neuromodulation in patient with chronic migraine. The study hypothesis to be tested is the mean reduction in mean monthly headache days between patients in treatment versus sham.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 22 years of age.
2. Have migraine onset at ≤ 50 years of age.
3. Have a history of migraine for ≥ 12 months prior to screening.
4. Have 15 - 26 headache days/month, among which ≥ 8 days has the features of probable migraine, and minimum of 2 headache-free days/month during the 28-day screening period.
5. Fulfill the criteria for chronic migraine (CM) during the 28-day screening period.
6. Have a diagnosis of refractory chronic migraine (RCM), who have inadequate response or no access to, or are intolerant, unwilling, or contraindicated to Onabotulinum toxin A (Botox) therapy, and One of the medications that belong to Calcitonin Gene Related Peptide Monoclonal antibodies (CGRP) therapy or CGRP antagonist therapy.
7. Maintain a stable use of preventive(s) migraine medication for ≥ 3 months before screening. Subjects receiving OnabotunlinumtoxinA must stop therapy ≥ 3 months prior to screening visit.
8. Demonstrate ≥ 80% compliance with the headache diary during the screening period by entering headache data on a minimum of 22 out of 28 days.
9. Be willing and able to comply with all study procedures and return to the clinic for the follow-up evaluation, as specified in this protocol.
10. Be able to give voluntary, written informed consent to participate in this study.

Exclusion Criteria:

1. Type of headache or migraine other than RCM including the following:

   1. Post-traumatic headache (e.g., battlefield, accidents, etc.).
   2. Regular intake of opioids (including codeine) of ≥ 8 days in the past 3 months and during the 28-day screening/baseline phase and cannot be accounted for by another diagnosis.
   3. Regular intake of Barbiturates for ≥ 5 days/month in the past 3 months and during the 28-day screening/baseline phase and cannot be accounted for by another diagnosis.
   4. Report experiencing unremitting, continuous headaches with no relief.
   5. Have new daily persistent headache (NDPH) defined by iCHD-3 as persistent headache, daily from its onset, which is clearly remembered. The pain lacks characteristic features and may be migraine-like or tension-type like or have elements of both with a CM subtype.
2. History of treatments that could confound the results of the study

   1. Previously implanted neurostimulator to stimulate the greater occipital and/or supraorbital nerves to treat headache.
   2. Have received onabotulinumtoxinA (Botox) for any other medical or cosmetic reasons requiring injections in the head, face, or neck within 3 months prior to screening.
3. Have had any cervical radiofrequency ablation within 12 months.
4. Subjects with recent brain or facial trauma occurring less than 3 months prior to the Baseline Visit.
5. Subjects that may have received sequential multi-day in-patient parenteral infusion for the treatment of a migraine condition (e.g., status migrainosus) within the previous 2 weeks of the initiation of diary screening phase.
6. Subjects with any metallic implant located in the head including CSF shunt and surgical clip above the shoulder line (excluding dental implants).
7. Subject has other implanted electrical stimulation device(s) including:

   1. Cardiac pacemakers or defibrillators
   2. Cochlear implant
   3. Intrathecal pumps
   4. Spinal cord stimulator
   5. Other stimulator device
8. Use of nerve blocks, acupuncture, neurostimulation and/or transcranial magnetic stimulation) for migraine within 3 months prior to screening and after receiving implant system.
9. Any pre-existing or requirement of emergent surgery/procedure that may interfere or confound the results of the study.
10. Any known requirement for an MRI scan subsequent to implant of the neurostimulator.
11. Current or history of following comorbidities:

    1. Clinically significant psychiatric illnesses, including suicide attempt, or suicidal ideation with a specific plan in the past 2 years.
    2. Cancer in the past 5 years, except for appropriately treated nonmelanoma skin carcinoma.
    3. Have a current diagnosis or condition that presents excess risk for performing the procedure, as determined clinically by the Investigator.
    4. Substance use disorder of at least moderate severe for substances such as; alcohol, recreational marijuana, or illicit drugs during the past 2 years.
12. Unable to participate or successfully complete the study, in the opinion of the investigator.
13. Anatomy not suitable for placement of the study device.
14. Are currently a study center or Sponsor employee who is directly involved in the study or the relative of such an employee.
15. Pregnant or lactating female or planning a pregnancy during participation in the study.
16. Patient with life expectancy of less than 1.5 years.
17. Currently participating in or planning to participate in other investigational drug or device studies that may interfere or confound the results of the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Headache Days | 12-weeks
  Mean monthly headache days

CONTACTS AND LOCATIONS:
Overall Officials: Brian Grosberg, MD, Principal Investigator — Hartford Headache Center; Samer Narouze, MD, Principal Investigator — University Hospitals
Locations (23):
- United States (20):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UC San Diego Health, La Jolla, California
  - Neurovations, Napa, California
  - Barolat Neuroscience, Denver, Colorado
  - Ayer Neuroscience Institute Headache Center, Hartford, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - Vista Clinical Research and Summit Spine & Joint, Newnan, Georgia
  - Synergy Headache Center & University of Illiniois Chicago, Chicago, Illinois
  - iSpine Clinics, Chaska, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Dent Neurologic Institute, Amherst, New York
  - Northwell Health Physician Partners, New York, New York
  - Montefiore Health, New York, New York
  - Queen City Clinical Research, Charlotte, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Argires Marotti Neurological Associates, Lancaster, Pennsylvania
  - Jefferson Headache Center, Philadelphia, Pennsylvania
  - Texas Neurology, Dallas, Texas
- Australia (3):
  - Genesis Research Services, Broadmeadow, New South Wales
  - CerCare, Wayville, South Australia
  - Monash House Research Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No